CLINICAL TRIAL: NCT07141732
Title: Pilot Prospective Single-center Non-comparative Study: Combined Treatment of Patients With Newly Diagnosed Glioblastoma Using the Xoft® Axxent® Electronic Brachytherapy (eBx®) System for Intraoperative Balloon Electronic Brachytherapy
Brief Title: Combined Treatment of Patients With Newly Diagnosed Glioblastoma Using the Xoft® Axxent® Electronic Brachytherapy (eBx®) System for Intraoperative Balloon Electronic Brachytherapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Joint Stock Company European Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1
Record Dates: First submitted 2025-08-15; First posted 2025-08-26 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; INTRAOPERATIVE BRACHYTHERAPY; RADIOTHERAPY
MeSH Terms: conditions — Glioblastoma | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glioblastoma (Experimental): Fifteen patients (male and female) with newly diagnosed glioblastoma who meet the inclusion/exclusion criteria (see below for details)
  Interventions: Biological: Resection of newly diagnosed glioblastoma combined with intraoperative balloon electronic brachytherapy using the Xoft® Axxent® Electronic Brachytherapy (eBx®) System

INTERVENTIONS:
Biological: Resection of newly diagnosed glioblastoma combined with intraoperative balloon electronic brachytherapy using the Xoft® Axxent® Electronic Brachytherapy (eBx®) System — The Elekta Xoft® Axxent® Electronic Brachytherapy (eBx®) System is a device that delivers high-dose-rate radiation. It is designed for use with Axxent applicators to treat neoplastic tumors inside or on the body surface where radiation therapy is indicated. The Axxent System and its applicators were cleared by the FDA under 510(k) submissions K050843, K072683, K090914, and K122951. The Russian Federation medical device registration certificate (No. RZN 2015/2593) was obtained on April 17, 2015.

SUMMARY:
Glioblastoma is the most aggressive primary brain tumor due to its highly infiltrative growth pattern, strong proliferative potential, and multiple mechanisms of resistance to treatment . Based on results from multicenter studies, English oncologist Roger Stupp proposed in 2005 a new treatment approach involving initial tumor resection followed by conformal external beam radiation therapy combined with temozolomide, plus subsequent cycles of monochemotherapy with this drug. This approach extended median survival by only 2 months, yet remains the standard of care due to lack of better alternatives. Consequently, recent protocols for malignant CNS tumors in Russia and internationally recommend prioritizing clinical trial enrollment over "standard" treatment.

Numerous studies demonstrate that the extent of resection of contrast-enhancing GB volume on MRI positively correlates with progression-free and overall survival. This is explained by the fact that adjuvant chemoradiation methods and the body's immune responses show efficacy only with small residual tumor volumes. The interval between surgery and adjuvant therapy negatively correlates with survival outcomes, potentially because the mitotic cycle of GB stem cells lasts only 24 hours. From this perspective, intraoperative radiation therapy (IORT) may improve treatment results.

Attempts to use various IORT technologies for malignant brain gliomas span several decades. Some studies reported better survival with IORT compared to controls, but most involved small patient groups without reliable resection control or dosimetric assessment due to technological limitations.

Early IORT methods used bulky linear accelerators producing high-energy electron beams. With portable systems, renewed interest emerged first in breast cancer, then neurosurgery. Neuroimaging and software now enable precise treatment planning. Bensaleh S. et al. evaluated balloon brachytherapy (MammoSite®) for early breast cancer in 2009. The device featured a dual-lumen catheter with a balloon inserted into the resection cavity. After contrast inflation and CT planning, 192Ir delivered 34 Gy in 10 fractions over 5 days to 1 cm depth. While comparable to conventional radiotherapy in 3-5 year survival, the 16% infection rate from prolonged implantation was a major drawback.

A case report described using a similar breast cancer system (Contura balloon applicator) for recurrent malignant glioma in a 47-year-old patient. A single 20 Gy fraction showed no complications at 6-month follow-up.

The Zeiss INTRABEAM system uses a miniature 50 kV linear accelerator with rigid spherical applicators producing low-energy x-rays for high surface doses with limited penetration. The 2018 INTRAGO phase I/II trial by Giordano et al. evaluated dose escalation (20→40 Gy) in 15 newly diagnosed GB patients. No complications (wound healing issues, bleeding, ischemia, or radionecrosis requiring surgery) occurred. Median PFS was 17.7 months (95% CI 9.7-25.9) in protocol-compliant patients, with distant progression remaining challenging.

A recent advancement is electronic brachytherapy using the Xoft Axxent eBx System, combining a 50 kV x-ray source with a silicone balloon applicator conforming to resection cavities. Initially successful in breast and gynecologic cancers, its application expanded to neuro-oncology.

In 2016, the European Medical Center (EMC) initiated a pilot study using Axxent eBx for recurrent GB post-standard chemoradiation. Twenty-nine patients received 20 Gy to the balloon surface after maximal safe resection. Median OS was 28.7 months (range 14-104) from first surgery. In patients with ≤2.5 cm³ residual tumor (n=16), median local PFS was 14.5 months (8-94), with 6- and 12-month PFS rates of 68.9% and 31% respectively. One grade 3 radionecrosis case occurred (CTCAE), with no infections or CSF leaks.

Study Rationale:

* Demonstrated survival benefits with gross-total resection of contrast-enhancing tumor
* Negative survival impact of delayed adjuvant therapy initiation
* Promising preliminary results of resection plus electronic brachytherapy in recurrent GB from EMC research This is a pilot, prospective, single-center, non-comparative study. Patients (N=15) with newly diagnosed glioblastoma will undergo intraoperative balloon-based electronic brachytherapy (IOBT) using the Xoft® Axxent® eBx® System immediately following gross total resection of the contrast-enhancing tumor. A single fractional dose of 20 Gy will be delivered to the balloon surface.

Subsequently, patients will receive standard chemoradiotherapy according to the Stupp protocol (2005):

* Concurrent phase (initiated 2-4 weeks postoperatively):

  * Radiotherapy: Conformal external beam radiation therapy (EBRT) to a total dose of 60 Gy (2 Gy/fraction over 6 weeks).
  * Chemotherapy: Daily oral temozolomide (75 mg/m²) during EBRT.
* Adjuvant phase:

  * Monotherapy: 6-12 cycles (6-12 months) of adjuvant temozolomide (150-200 mg/m², days 1-5 of each 2

ELIGIBILITY:
Inclusion Criteria:

* The subject's age must be ≥ 40 years but not older than 75 years.
* The subject's Karnofsky Performance Status (KPS) must be ≥ 70%.
* The subject is willing and able to independently provide informed consent for participation in the study.
* The subject has been newly diagnosed with glioblastoma (GB) based on preoperative neuroimaging (contrast-enhanced brain MRI ± amino acid-based PET/CT) and confirmed by intraoperative histopathological examination of the tumor.
* Total or near-total resection of the contrast-enhancing tumor portion is feasible.
* The expected post-resection cavity size must allow placement of the Axxent Xoft eBx balloon applicator system.
* Women of childbearing potential must have a negative pregnancy test within 7 days before treatment initiation.
* The subject must have a complete blood count (CBC) with or without differential within 7 days before study enrollment, demonstrating adequate bone marrow function:

  * Absolute neutrophil count (ANC) ≥ 1500 cells/mm³
  * Platelets ≥ 75,000 cells/mm³
  * Hemoglobin ≥ 10.0 g/dL
* The subject must undergo kidney and liver function tests within 7 days before study enrollment, with the following required parameters:

  * Total bilirubin ≤ 2.0 mg/dL, and AST ≤ 2.5 × upper limit of normal (ULN)
  * Serum creatinine ≤ 1.8 mg/dL within 14 days before enrollment.
* The subject's urine protein levels must meet the following criteria within 14 days before enrollment:

  * Urine protein-to-creatinine ratio (UPCR) < 1.0, OR
  * Dipstick urinalysis ≤ 2+ proteinuria (if > 2+, a 24-hour urine collection must show ≤ 1 g protein/24h).
* Patients on anticoagulant therapy (e.g., warfarin or low-molecular-weight heparin) must meet all of the following:

  * No active bleeding or high-risk bleeding conditions (e.g., tumor involving major vessels or varices).
  * Stable INR (typically 2-3) on oral anticoagulants OR stable dose of LMWH for ≥ 14 days before enrollment.

Exclusion Criteria:

* Multicentric/multifocal glioblastoma growth.
* Infratentorial or leptomeningeal tumor spread.
* Recurrent/progressive glioblastoma.
* Prior cranial radiation therapy.
* Glioblastoma located in or near (≤ 10 mm from) critical brain structures, preventing adequate radiation dose delivery.
* Contrast-enhancing tumor diameter > 6 cm.
* Active or prior malignancy (except adequately treated non-melanoma skin cancer or carcinoma in situ).
* Other intracranial neoplasms (current or history).
* Pregnancy, lactation, or unwillingness to use effective contraception (for women of childbearing potential or sexually active men).
* Contraindications to MRI (with or without gadolinium).
* Non-removable or clinically inoperable cardiac pacemaker/device.
* Contraindications to general anesthesia.
* Concurrent participation in another clinical trial.
* Severe comorbidities, including:

  * Unstable angina or congestive heart failure requiring hospitalization (within 6 months).
  * Transmural myocardial infarction (within 6 months).
  * Stroke or transient ischemic attack (within 6 months).
  * Significant vascular disease (aortic/peripheral).
  * Active venous/arterial thromboembolism.
  * Acute bacterial/fungal infection requiring IV antibiotics.
  * COPD exacerbation or respiratory disease interfering with protocol therapy.
  * Liver failure causing jaundice/coagulopathy.
* Positive serology for HIV, HBV, HCV, or syphilis.
* Grade ≥ 3 hemorrhage (CTCAE v5.0) within 30 days before enrollment.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint - Overall Survival (OS) of patients | Overall Survival (OS) of patients, assessed at 16 and 36 months from the start of treatment per the study protocol. Units of Measure is month.

SECONDARY OUTCOMES:
• Local Progression-Free Survival (L-PFS) • Distant Progression-Free Survival (D-PFS) | Assessed at 16 and 36 months from treatment initiation. Units of Measure is month.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksey Krivoshapkin, Professor M.D., Principal Investigator — Joint-Stock Company European Medical Center; Alexey Gaitan, Candidate of Medical Sciences, Principal Investigator — Joint-Stock Company European Medical Center
Locations (1):
- Joint-Stock Company European Medical Center, Moscow, Moscow, Russia